CLINICAL TRIAL: NCT06516133
Title: Artificial Intelligence Empowered Online Adaptive Radiotherapy Versus Conventional Radiotherapy in Non-metastatic Nasopharyngeal Carcinoma: an Open-label, Non-inferiority, Multicentre, Randomised Phase 3 Trial
Brief Title: Online Adaptive Radiotherapy for Nasopharyngeal Carcinoma
Acronym: OART
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, YingSun, Principal Investigator, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SL-B2023-685-02
Record Dates: First submitted 2023-12-27; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma; Online adaptive radiotherapy; Smaller PTV margin
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Radiotherapy, Intensity-Modulated; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional radiotherapy with conventional margins w or w/o chemotherapy (Active Comparator): Complete the full course of radiotherapy using the original treatment plan. PTV margin: 3mm.
  Interventions: Radiation: Intensity modulated radiation therapy (IMRT) with conventional planning target volume (PTV) margin and without online adaptive radiotherapy; Drug: Chemotherapy
- Radiotherapy with smaller margin and online adaptive radiotherapy w or w/o chemotherapy (Experimental): Throughout the course of radiotherapy, the treatment plan is adjusted online based on the anatomical and dosimetric changes in the target volumes and organs at risk of the patients.
  PTV margin: smaller.
  Interventions: Radiation: Intensity modulated radiation therapy (IMRT) with smaller planning target volume (PTV) margin and online adaptive radiotherapy; Drug: Chemotherapy

INTERVENTIONS:
Radiation: Intensity modulated radiation therapy (IMRT) with conventional planning target volume (PTV) margin and without online adaptive radiotherapy — Radiation: Complete the full course of radiotherapy using the original treatment plan.
  Planning target volume (PTV) margin: 3mm;
  Arms: Conventional radiotherapy with conventional margins w or w/o chemotherapy
Drug: Chemotherapy — Chemotherapy: If given, platinum-based.
  Arms: Conventional radiotherapy with conventional margins w or w/o chemotherapy
Radiation: Intensity modulated radiation therapy (IMRT) with smaller planning target volume (PTV) margin and online adaptive radiotherapy — Radiation: During the course of radiotherapy, the treatment plan is adjusted online based on the anatomical and dosimetric changes in the target volumes and organs at risk of patients.
  planning target volume (PTV) margin: smaller.
  Arms: Radiotherapy with smaller margin and online adaptive radiotherapy w or w/o chemotherapy
Drug: Chemotherapy — Chemotherapy: If given, platinum-based
  Arms: Radiotherapy with smaller margin and online adaptive radiotherapy w or w/o chemotherapy

SUMMARY:
In this multicenter, prospective, randomized, controlled, non-inferiority Phase III clinical trial, treatment-naïve patients with nasopharyngeal carcinoma (NPC) without metastasis will be enrolled for curative radiotherapy. The participants will be randomly assigned to two groups. The experimental group will receive online adaptive radiotherapy (ART) during the radiotherapy process, with a smaller PTV margin, while the control group will use original treatment plan during full-course radiotherapy, with a PTV margin of 3 mm. The study aims to compare the survival, adverse events, and quality of survival between the two groups, with the primary endpoint being the locoregional recurrence-free survival rate. The main objective is to determine the role of online ART in nasopharyngeal carcinoma, elucidating its potential to alleviate radiation toxicity in patients while ensuring treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed nasopharyngeal carcinoma confirmed by pathology, with a histological classification of non-keratinizing carcinoma (according to the World Health Organization, WHO), pathological classification.
2. No evidence of distant metastasis (M0).
3. Age between 18 and 70 years.
4. Eastern Cooperative Oncology Group (ECOG) performance status score:0-1.
5. Undergoing radical intensity-modulated radiation therapy (IMRT).
6. No claustrophobia and able to remain in a fixed position for at least 30 minutes
7. Patients must be informed of the main content of this study, sign an informed consent form, and be willing and able to comply with the treatment, follow-up plan, laboratory tests, and other requirements specified in the study protocol.

Exclusion Criteria:

1. Histological types include squamous cell carcinoma or basal cell carcinoma.
2. Radiation therapy intended for palliative care.
3. History of malignant tumors, excluding adequately treated basal cell carcinoma, squamous cell carcinoma, and cervical intraepithelial neoplasia.
4. Pregnant or lactating women (women of childbearing age should undergo pregnancy testing; effective contraception should be emphasized during treatment.
5. Previous radical radiotherapy for nasopharyngeal cancer.
6. Primary and neck metastatic lesions treated with chemotherapy or surgery.
7. Presence of other serious underlying diseases that may pose a greater risk or affect compliance with the trial. Examples include unstable cardiac diseases requiring treatment, renal diseases, chronic hepatitis, poorly controlled diabetes (fasting blood glucose > 1.5×ULN), and psychiatric disorders.
8. Initial assessment of treatment efficacy more than 120 days after the end of radiotherapy.
9. Inability to undergo enhanced magnetic resonance imaging due to contrast agent allergies, claustrophobia.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 494 (Estimated)
Dates: Start 2024-05-17 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Locoregional recurrence-free survival | 3-year
  locoregional progression free survival

SECONDARY OUTCOMES:
Overall survival | 3-year
  overall survival
Distant metastasis free survival | 3-year
  Distant metastasis free survival
Rate of acute radiation-induced events according to Common Terminology Criteria for Adverse Events (CTCAE 5.0) | 3 months
  Acute radiation-induced events. The minimum and maximum values are 0 and 5 respectively. The higher scores mean a worse outcome.
Rate of late radiation-induced events according to Common Terminology Criteria for Adverse Events (CTCAE 5.0). | 3-year
  Late radiation-induced events. The minimum and maximum values are 0 and 5 respectively. The higher scores mean a worse outcome.
European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Head and Neck 35 Version 1.0 (EORTC QLQ-HN35 V1.0) | From baseline to 3 years post-radiotherapy
  The minimum and maximum values are 0 and 4 respectively. The higher scores mean a worse outcome.
and National Cancer Institute Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events Version 1.0 (NCI-PRO-CTCAE V1.0.) | From baseline to 3 years post-radiotherapy
  The minimum and maximum values are 0 and 5 respectively. The higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No